CLINICAL TRIAL: NCT03428815
Title: Effects of Temperature Control Liner Materials on Long-Term Outcomes of Prothesis Use
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Pandemic response invalidated long-term outcome data collection
Sponsor: Goeran Fiedler (Other)
Collaborators: Widener University (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Goeran Fiedler, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO17090574; W81XWH-16-OPORP-PORA (Other Grant/Funding Number: US Dept of Defense)
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Results first posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Artificial Limbs; Skin Diseases
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PCM liner (Experimental): Willowwood Smart Temp Liner
  Interventions: Device: Prosthesis suspension liner
- regular liner (Active Comparator): User's regular prescribed liner
  Interventions: Device: Prosthesis suspension liner

INTERVENTIONS:
Device: Prosthesis suspension liner — Liners out of phase change material will be fitted

SUMMARY:
This clinical trial will compare how many days per year people with lower limb prosthesis do not wear their prosthesis when fitted with a conventional liner and a liner made with phase change materials.

DETAILED DESCRIPTION:
Background: The proposed work will generate evidence-based practice guidance for temperature control liner technologies and allow providers to optimize care to Service members and Veterans with limb loss. Sizeable numbers of Service members and Veterans live with limb loss, mostly due to traumatic musculoskeletal injury. Addressing the resulting functional deficit with prostheses increases the risk for secondary conditions such as pressure sores, impaired blood perfusion, and injuries from accidental falls. Any of those occurrences can render the prosthesis temporarily useless, making it challenging for users to engage in many activities of daily life, including work, exercise, and social participation. Many of the described issues originate at the interface between residual limb and prosthetic socket, where the objectives of sufficient weight distribution and suspension are conflicting with the necessity to facilitate heat exchange and limit contact pressure and friction.

Recently, prosthesis liners that contain phase-change material have become commercially available, holding the promise that the micro climate at the interface between the residual limb skin and the prosthetic socket can be regulated to reduce the users' tendency to sweat. Preliminary studies on these liners indicate that the socket temperatures inside the socket stayed lower and rose slower than in conventional liners. However, the clinical relevance of those findings remains unclear. While (perceived) socket comfort is certainly an important criterion in prosthesis fitting, it may be claimed that only tangible functional benefits are of concern.

Objective/Hypothesis: The purpose of this study is to investigate whether longer (6+ months) periods of use of phase-change material based temperature control liners have clinically meaningful effects.

It is hypothesized that use of phase-change material infused liners will improve prosthesis utilization (measured in days of prostheses use per time), physical performance (measured by 2-minute walk test), and self-reported prosthesis related quality of life (assessed by questionnaire). The research follows the rationale that lower and steadier skin temperatures should result in reduced sweat, friction, skin damage, and prosthesis abandonment. This would encourage users to wear their prosthesis for longer periods of time and for an expanded array of purposes, thus increasing their ability to ambulate and to engage in a greater variety of activities.

Specific Aims:

1. To compare phase-change material liners to conventional liners with regard to activity and participation
2. To quantify the effect of phase-change material liners on prosthesis related quality of life and physical performance over time
3. To investigate the relationship between perceived benefits of phase-change material liners and patient-centric outcomes

Study Design: The proposed study will utilize a double-blind longitudinal cross-over research design. A sample of trans-tibial prosthesis users will be wearing their regular gel or silicone liners for six months and phase-change material liners for another six months in a randomized sequence. Their prostheses will be equipped with activity monitors, and participants will be asked to maintain a record of days when they could not wear their prosthesis due to any perceived issues with their residual limb or socket fit. In 1.5-month intervals, subjects' activity, physical performance, and overall prosthesis assessment will be recorded using standardized methods.

ELIGIBILITY:
Inclusion Criteria:

* use of a prosthesis with liner suspension,
* at least one year of prosthesis use,
* a well-fitting socket,
* a matured residual limb (stable limb volume) that has not required socket modifications in the previous year,
* the ability to walk with the prosthesis outdoors without notable limitations (K-Level 3),
* stable weight,
* absence of acute medical conditions that would temporarily affect the ability to use prostheses.

Exclusion Criteria:

* use of a non-standard liner size,
* current use of a PCM liner as the regular suspension system,
* known allergies against liner materials,
* any inability to understand the protocol and to comply with the associated tasks, such as maintaining a log of days when the prosthesis could not be used.
* anticipated provision of a new prosthesis or extended (longer than one month) absences from the region during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bakery Square MSPO labs, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data may be shared in the future

REFERENCES:
- [Derived] Fiedler G, Singh A, Zhang X. Effect of temperature-control liner materials on long-term outcomes of lower limb prosthesis use: a randomized controlled trial protocol. Trials. 2020 Jan 10;21(1):61. doi: 10.1186/s13063-019-3920-4. PMID 31924257
- See also: Details on the PLUS-M mobility scale used for baseline assessment — http://plus-m.org/about.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Six participants did not start the protocol: Four had an incompatibility of study liners with their existing socket prosthesis, one had an unrelated health issue, and one was unreachable after enrollment.
Groups:
- First PCM Liner, Then Regular Liner: Prosthesis suspension liner: Liners out of phase change material (Willowwood Smart Temp Liner) are fitted first. After 6 months they are exchanged against a set of regular liners
- First Regular Liner, Then PCM Liner: Prosthesis suspension liner: Participants' regular liners are fitted first. After 6 months they are exchanged against a set of phase change material liners (Willowwood Smart Temp Liner)
Period: Overall Study
Arm/Group | First PCM Liner, Then Regular Liner | First Regular Liner, Then PCM Liner
Started | 17 | 19
Completed | 7 | 14
Not Completed | 10 | 5
Not completed — Lost to Follow-up | 2 | 2
Not completed — suspension of study activities due to Covid-19 pandemic | 5 | 2
Not completed — Intermittent fitting issues that affected reliability of data | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCM Liner | Regular Liner | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (13) | 59 (11) | 57 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 15 | 13 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17 | 19 | 36
Height [Mean (Standard Deviation); unit: cm] | 181 (7) | 175 (11) | 178 (10)
Weight [Mean (Standard Deviation); unit: kg] | 97 (23) | 99 (24) | 98 (23)
Years since limb loss [Mean (Standard Deviation); unit: years] | 8 (7) | 10 (12) | 9 (10)
Mobility score (z-score, PLUS-M) [Mean (Standard Deviation); unit: units on a scale] — Prosthetic Limb User Survey-Mobility (PLUS-M) is a survey instrument that uses a set of standardized calibrated questions. The z-score indicates the respondent's mobility score with respect to the normal distribution of the general lower limb prosthesis user population. This distribution has a mean value of 50 and a standard deviation of 10. Higher scores indicate greater levels of mobility.
  units on a scale | 57 (6) | 55 (8) | 56 (7)

OUTCOME MEASURES:

1. Primary Outcome: Days Without Prosthesis
Description: Days with less than 10% of prosthesis steps than the individual's daily average across the study period. Days without prosthesis are prorated to a full year (365 days) for comparison purposes.
Time Frame: 6 months
Population: only participants with data from both interventions (cross-over design) was included
Measure: Mean (Full Range); unit: prorated days per year
Arm/Group | PCM Liner | Regular Liner
Number analyzed (Participants) | 21 | 21
prorated days per year | 17 [0 to 21] | 19 [0 to 35]

2. Secondary Outcome: Average Daily Step Count
Description: A participant's daily step counts were averaged across days with prosthesis use across each intervention period
Time Frame: 6 months per intervention
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | PCM Liner | Regular Liner
Number analyzed (Participants) | 21 | 21
steps per day | 2053 (1249) | 2117 (1176)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Of the 42 participants that were enrolled (i.e., screened and signed the consent form), 36 received liners (19 received the PCM liner first and 17 received the regular liner first). After some attrition, 16 of the first group received the regular liner and ten of the second group received the PCM liner. Therefore, a total of 29 participants were exposed to the PCM liner and 33 to the regular liner during the study.
Arm/Group | PCM Liner | Regular Liner
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/33
Other Adverse Events (participants affected / at risk) | 1/29 | 0/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCM Liner (N=29) | Regular Liner (N=33)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Liner damage that caused skin irritation was determined to be normal wear and tear

LIMITATIONS AND CAVEATS:
Covid-19 pandemic invalidated assumptions about the representativeness of daily step counts and led to early termination of enrollment and ongoing data collection. The remaining sample size was insufficient for the planned analyses beyond descriptive statistics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT03428815/Prot_SAP_001.pdf